CLINICAL TRIAL: NCT01077362
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Ustekinumab, a Fully Human Anti-IL-12/23p40 Monoclonal Antibody, Administered Subcutaneously, in Subjects With Active Psoriatic Arthritis Including Those Previously Treated With Biologic Anti-TNFalpha Agent(s)
Brief Title: A Study of the Safety and Efficacy of Ustekinumab in Patients With Psoriatic Arthritis With and Without Prior Exposure to Anti-TNF Agents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016483; CNTO1275PSA3002 (Other: Janssen Research & Development, LLC); 2009-012265-60 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Arthritis, Psoriatic
Keywords: Ustekinumab; CNTO 1275; Stelara; Psoriatic Arthritis; Psoriasis; TNF alpha
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Experimental): Participants will receive subcutaneous (SC) injections of placebo at Weeks 0, 4, 16, and 20. At Week 24 participants will cross over to receive SC injections of ustekinumab 45 mg at Weeks 24 and 28 and every 12 weeks thereafter with the last dose at Week 40. If early escape, SC injections of 45 mg ustekinumab will be given at Weeks 16, 20, and 28 and every 12 weeks thereafter with the last dose at Week 40. For participants entering early escape, a SC placebo injection will be given at Week 24 to maintain the blind.
  Interventions: Drug: placebo
- Ustekinumab 45 mg (Experimental): Participants will receive SC injections of ustekinumab 45 mg at Weeks 0 and 4 and every 12 weeks thereafter with the last dose at Week 40. If early escape, SC injections of 90 mg ustekinumab will be given at Week 16 and every 12 weeks thereafter with the last dose at Week 40. Participants will receive SC injections of placebo at Weeks 20 and 24 to maintain the blind.
  Interventions: Drug: placebo; Drug: ustekinumab 45 mg; Drug: ustekinumab 90 mg
- Ustekinumab 90 mg (Experimental): Participants will receive SC injections of ustekinumab 90 mg at Weeks 0 and 4 and every 12 weeks thereafter with the last dose at Week 40. If early escape, the same dosage schedule will continue. Participants will receive SC injections of placebo at Weeks 20 and 24 to maintain the blind.
  Interventions: Drug: placebo; Drug: ustekinumab 90 mg

INTERVENTIONS:
Drug: placebo — SC injections
Drug: ustekinumab 45 mg — SC injections
  Arms: Ustekinumab 45 mg
Drug: ustekinumab 90 mg — SC injections
  Arms: Ustekinumab 45 mg; Ustekinumab 90 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy (improvement of signs and symptoms) and safety of ustekinumab in patients with psoriatic arthritis.

DETAILED DESCRIPTION:
This study is a randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), parallel-group, multicenter study to evaluate the effectiveness and safety of ustekinumab compared to placebo in the treatment of patients with active psoriatic arthritis who have or are currently receiving treatment with a disease-modifying antirheumatic drug (DMARD) and/or a nonsteroidal anti-inflammatory drug (NSAID), including those who have previously received anti-tumor necrosis factor (anti-TNF) agents [(examples are infliximab (Remicade), etanercept (Enbrel), adalimumab (Humira)]. The primary effectiveness endpoint will be measured by the reduction in signs and symptoms of arthritis, as defined by 20% improvement from baseline in American College of Rheumatology (ACR) measurements of arthritis at Week 24. The study will additionally look at higher levels of joint improvement (ie, 50% or 70% improvement from baseline) and improvement in activity and quality of life, as well as the impact of ustekinumab on psoriatic skin lesions. Safety assessments will be performed throughout the study and include obtaining and evaluating laboratory tests, vital signs (eg, blood pressure) and the occurrence and severity of adverse events (side effects). Patients will be assigned to one of three treatment groups. Patients will receive either 45 mg ustekinumab, 90 mg ustekinumab, or placebo at Weeks 0, 4 and every 12 weeks until Week 40. Patients who do not have >=5% improvement in their disease (tender and swollen joints) at Week 16 may be eligible to receive an increase or change to their ustekinumab dosage. Ustekinumab 45 mg, 90 mg, or placebo subcutaneous injections at Weeks 0 and 4 followed by every-12-week dosing with the last dose at Week 40. Early escape possibility at Week 16. Patients randomized to placebo will crossover to receive ustekinumab at Weeks 24 and 28 followed by every-12-week dosing with the last dose at Week 40. Expected duration of exposure to study agent including follow up for safety is 60 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have had a documented diagnosis of psoriatic arthritis (PsA) at least 6 months
* Have a diagnosis of active PsA at the time of entry into the study with at least 5 tender and 5 swollen joints at baseline
* May have previously received at least 8 weeks of etanercept, adalimumab, golimumab or certolizumab pegol or at least 14 weeks of infliximab or proven inability to tolerate anti-TNF therapy for 8-14 weeks
* If the patient is using methotrexate, they should have started treatment at a dose not to exceed 25 mg/week at least 3 months prior to the beginning of the study and should have no serious toxic side effects attributable to methotrexate

Exclusion Criteria:

* Have other inflammatory diseases, including but not limited to rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, or Lyme disease
* Have used any therapeutic agent targeted at reducing IL-12 or IL-23, including but not limited to ustekinumab and ABT-874
* Have used infliximab, golimumab or certolizumab pegol within 12 weeks of first study drug injection, or etanercept or adalimumab within 8 weeks of first study drug injection
* Have a medical history of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis, prior to screening
* Have any known malignancy or have a history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or cervical carcinoma in situ that has been treated with no evidence of recurrence, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years of the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (80):
- United States (25):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Los Angeles, California
  - San Diego, California
  - Denver, Colorado
  - Trumbull, Connecticut
  - Tampa, Florida
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - Wheaton, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Edina, Minnesota
  - Clayton, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Freehold, New Jersey
  - Orchard Park, New York
  - Rochester, New York
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - West Reading, Pennsylvania
  - Dallas, Texas
- Austria (3):
  - Graz
  - Sankt Pölten
  - Vienna
- Canada (16):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - Barrie, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - North Bay, Ontario
  - Saint Catherines, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Trois-Rivières, Quebec
- France (6):
  - Bordeaux
  - Chambray-lès-Tours
  - Créteil
  - Lille
  - Paris
  - Toulouse
- Germany (6):
  - Berlin
  - Cologne
  - Erlangen
  - Hamburg
  - Herne
  - München
- Hungary (3):
  - Debrecen
  - Szombathely
  - Veszprém
- Poland (4):
  - Bialystok
  - Bydgoszcz
  - Lublin
  - Warsaw
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Yekaterinburg
- Sweden (4):
  - Gothenburg
  - Malmo
  - Stockholm
  - Uppsala
- United Kingdom (10):
  - Cannock
  - Glasgow
  - London
  - Metropolitan Borough of Wirral
  - Newcastle upon Tyne
  - Salford
  - Sheffield
  - Southampton
  - Westcliff-on-Sea
  - Wigan

REFERENCES:
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Ustekinumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Oct;11(5):1413-1423. doi: 10.1007/s40744-024-00705-x. Epub 2024 Aug 9. PMID 39120848
- [Derived] Helliwell PS, Gladman DD, Chakravarty SD, Kafka S, Karyekar CS, You Y, Campbell K, Sweet K, Kavanaugh A, Gensler LS. Effects of ustekinumab on spondylitis-associated endpoints in TNFi-naive active psoriatic arthritis patients with physician-reported spondylitis: pooled results from two phase 3, randomised, controlled trials. RMD Open. 2020 Feb;6(1):e001149. doi: 10.1136/rmdopen-2019-001149. PMID 32209721
- [Derived] Siebert S, Sweet K, Dasgupta B, Campbell K, McInnes IB, Loza MJ. Responsiveness of Serum C-Reactive Protein, Interleukin-17A, and Interleukin-17F Levels to Ustekinumab in Psoriatic Arthritis: Lessons From Two Phase III, Multicenter, Double-Blind, Placebo-Controlled Trials. Arthritis Rheumatol. 2019 Oct;71(10):1660-1669. doi: 10.1002/art.40921. Epub 2019 Sep 3. PMID 31070869
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Rahman P, Puig L, Gottlieb AB, Kavanaugh A, McInnes IB, Ritchlin C, Li S, Wang Y, Song M, Mendelsohn A, Han C; PSUMMIT 1 and 2 Study Groups. Ustekinumab Treatment and Improvement of Physical Function and Health-Related Quality of Life in Patients With Psoriatic Arthritis. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1812-1822. doi: 10.1002/acr.23000. Epub 2016 Oct 21. PMID 27483458
- [Derived] Kavanaugh A, Puig L, Gottlieb AB, Ritchlin C, You Y, Li S, Song M, Randazzo B, Rahman P, McInnes IB. Efficacy and safety of ustekinumab in psoriatic arthritis patients with peripheral arthritis and physician-reported spondylitis: post-hoc analyses from two phase III, multicentre, double-blind, placebo-controlled studies (PSUMMIT-1/PSUMMIT-2). Ann Rheum Dis. 2016 Nov;75(11):1984-1988. doi: 10.1136/annrheumdis-2015-209068. Epub 2016 Apr 20. PMID 27098404

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received subcutaneous (SC) injections of placebo at Weeks 0, 4, 16, and 20. At Week 24 participants crossed over to receive SC injections of ustekinumab 45 mg at Weeks 24 and 28 and every 12 weeks thereafter with the last dose at Week 40. If early escape, SC injections of 45 mg ustekinumab were given at Weeks 16, 20, and 28 and every 12 weeks thereafter with the last dose at Week 40. For participants entering early escape, a SC placebo injection was given at Week 24 to maintain the blind.
- Ustekinumab 45 mg: Participants received SC injections of ustekinumab 45 mg at Weeks 0 and 4 and every 12 weeks thereafter with the last dose at Week 40. If early escape, SC injections of 90 mg ustekinumab were given at Week 16 and every 12 weeks thereafter with the last dose at Week 40. Participants received SC injections of placebo at Weeks 20 and 24 to maintain the blind.
- Ustekinumab 90 mg: Participants received SC injections of ustekinumab 90 mg at Weeks 0 and 4 and every 12 weeks thereafter with the last dose at Week 40. If early escape, the same dosage schedule continued. Participants received SC injections of placebo at Weeks 20 and 24 to maintain the blind.
Period: Overall Study
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Started | 104 | 103 | 105
Completed | 73 | 84 | 81
Not Completed | 31 | 19 | 24
Not completed — Lack of Efficacy | 13 | 8 | 10
Not completed — Lost to Follow-up | 1 | 0 | 3
Not completed — Adverse Event | 12 | 7 | 4
Not completed — Withdrawal by Subject | 5 | 3 | 5
Not completed — Other | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | Total
Number analyzed (Participants) | 104 | 103 | 105 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (11.19) | 48 (11.21) | 48.2 (12.36) | 47.9 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 55 | 56 | 164
  Male | 51 | 48 | 49 | 148

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 24.
Description: An ACR 20 response is defined as a greater than or equal to 20 percent improvement from baseline in swollen (66 joints) and tender (68 joints) joint counts and greater than or equal to 20 percent improvement in 3 of the following 5 assessments: 1) Participant's assessment of pain by Visual Analog Scale (VAS) (0-10 cm), 2) Participant's global assessment of disease activity by VAS (0-10 cm), 3) Physician's global assessment of disease activity by VAS (0-10 cm) 4) Participant's assessment of physical function as measured by the "Disability Index of the Health Assessment Questionnaire" (HAQ-DI) (score of 0-3 in 8 functional areas) and 5) C reactive protein.
Time Frame: Week 24
Population: All participants randomly assigned to a treatment group were included in the efficacy analysis regardless of whether they received the assigned treatment. For early escape, data at or prior to Week 16 were carried forward through Week 24.
Measure: Number; unit: Percentage of participants
Groups:
- All Ustekinumab Combined: Participants who received SC injections of ustekinumab at any dose (45 mg and 90 mg) through Week 40.
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 104 | 103 | 105 | 208
Percentage of participants | 20.2 | 43.7 | 43.8 | 43.8
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

2. Secondary Outcome: Change From Baseline to Week 24 in the Disability Index Score as Measured With the "Disability Index of the Health Assessment Questionnaire" (HAQ-DI)
Description: HAQ-DI is 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 (no difficulty), to 3 (inability to perform a task in that area). The average score across the functional areas yields an overall HAQ-DI score which ranges from 0 (no disability) to 3 (completely disabled). In psoriatic arthritis, a decrease in score of 0.30 indicates clinically meaningful improvement.
Time Frame: Day 1 (Baseline) and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 104 | 103 | 105 | 208
Score on a scale | -0.03 (0.380) | -0.21 (0.461) | -0.22 (0.436) | -0.21 (0.447)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p = 0.002, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

3. Secondary Outcome: Percentage of Participants (With >= 3% Baseline Body Surface Area (BSA) Psoriatic Involvement) Who Achieved a Psoriasis Area and Severity Index 75 (PASI 75) Response at Week 24
Description: The PASI is a physician-administered assessment tool used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 (no disease) to 72 (maximal disease). A PASI 75 response is defined as greater than or equal to 75 percent improvement in PASI score from baseline.
Time Frame: Week 24
Population: All participants randomly assigned to a treatment group were included in the efficacy analysis regardless of whether they received the assigned treatment. For early escape, data at or prior to Week 16 were carried forward through Week 24. Only participants with >=3% baseline BSA psoriatic involvement were included in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 80 | 80 | 81 | 161
Percentage of participants | 5.0 | 51.3 | 55.6 | 53.4
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

4. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50 Response at Week 24
Description: An ACR 50 response is defined as a greater than or equal to 50 percent improvement from baseline in swollen (66 joints) and tender (68 joints) joint counts and greater than or equal to 50 percent improvement in 3 of the following 5 assessments: 1) Participant's assessment of pain by Visual Analog Scale (VAS) (0-10 cm), 2) Participant's global assessment of disease activity by VAS (0-10 cm), 3) Physician's global assessment of disease activity by VAS (0-10 cm) 4) Participant's assessment of physical function as measured by the "Disability Index of the Health Assessment Questionnaire" (HAQ-DI) (score of 0-3 in 8 functional areas) and 5) C reactive protein.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 104 | 103 | 105 | 208
Percentage of participants | 6.7 | 17.5 | 22.9 | 20.2
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p = 0.018, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p = 0.002, re-randomization test

5. Secondary Outcome: Change From Baseline to Week 24 in Total Modified Van Der Heijde-Sharp (vdH-S) Score for the Combined Radiographic Data From Studies CNTO1275PSA3001 and CNTO1275PSA3002
Description: The modified vdH-S score is a radiographic evaluation of hand and feet erosions and joint space narrowing (JSN) for 20 joints per hand and 6 joints per foot with a total score ranging from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher scores and positive score changes indicate more radiographic damage and radiographic progression, respectively. As per protocol, the analysis for this outcome measure used pooled data from 2 studies (CNTO1275PSA3001 and PSA3002) because initial power assumptions showed that 900 participants would be required to evaluate the impact of ustekinumab on structural damage (SD) progression. The 2 studies, (which had similar study designs and dosing regimens and differed only with regards to prior exposure to anti-TNFα therapies), were intended to independently measure efficacy in terms of signs, symptoms and physical function, while effects on SD progression would be provided from an integrated analysis.
Time Frame: Day 1 (Baseline) and Week 24
Population: Analysis included: (1) combined data from studies CNTO1275PSA3001 (NCT01009086) and CNTO1275PSA3002 (NCT01077362) and (2) all participants randomly assigned to a treatment group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 310 | 308 | 309 | 617
Score on a scale | 0.97 (3.852) | 0.40 (2.110) | 0.39 (2.403) | 0.40 (2.260)
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p = 0.017, re-randomization test
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p < 0.001, re-randomization test

6. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 70 Response at Week 24
Description: An ACR 70 response is defined as a greater than or equal to 70 percent improvement from baseline in swollen (66 joints) and tender (68 joints) joint counts and greater than or equal to 70 percent improvement in 3 of the following 5 assessments: 1) Participant's assessment of pain by Visual Analog Scale (VAS) (0-10 cm), 2) Participant's global assessment of disease activity by VAS (0-10 cm), 3) Physician's global assessment of disease activity by VAS (0-10 cm) 4) Participant's assessment of physical function as measured by the "Disability Index of the Health Assessment Questionnaire" (HAQ-DI) (score of 0-3 in 8 functional areas) and 5) C reactive protein.
Time Frame: Week 24
Population: All participants randomly assigned to a treatment group were included in the efficacy analysis regardless of whether they received the assigned treatment. For early escaped, data at or prior to Week 16 were carried forward through Week 24.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | All Ustekinumab Combined
Number analyzed (Participants) | 104 | 103 | 105 | 208
Percentage of participants | 2.9 | 6.8 | 8.6 | 7.7
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 45 mg; Test type: Superiority or Other; p = 0.171, re-randomization
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p = 0.060, re-randomization test
Statistical Analysis 3: Comparison: Placebo vs All Ustekinumab Combined; Test type: Superiority or Other; p = 0.094, re-randomization

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the study (60 weeks).
Description: The safety analysis included all participants who were randomly assigned to a treatment group and received at least one dose of study agent, either placebo or ustekinumab. One participant, in the ustekinumab 90 mg group, did not receive treatment and is excluded from the safety analysis set.
Groups:
- Placebo: Controlled Period: Adverse events which occurred during Weeks 0-16 (placebo-controlled period) in participants who were randomly assigned to placebo at Baseline.
- Ustekinumab 45 mg: Controlled Period: Adverse events which occurred during Weeks 0-16 (placebo-controlled period) in participants who were randomly assigned to ustekinumab 45 mg at Baseline.
- Ustekinumab 90 mg: Controlled Period: Adverse events which occurred during Weeks 0-16 (placebo-controlled period) in participants who were randomly assigned to ustekinumab 90 mg at Baseline.
- Placebo: Weeks 16-24: Adverse events which occurred during Weeks 16-24 in participants who were randomly assigned to placebo at Baseline and did not early escape at Week 16.
- Placebo -> Ustekinumab 45 mg: Weeks 16-60: Adverse events which occurred (1) during Weeks 16-60 in participants randomly assigned to placebo at Baseline and who early escaped to ustekinumab 45 mg at Week 16 and (2) during Weeks 24-60 in participants randomly assigned to placebo at Baseline and who crossed over to ustekinumab 45 mg at Week 24.
- Ustekinumab 45 mg: Weeks 16-60: Adverse events which occurred during Weeks 16-60 in participants who were randomly assigned to ustekinumab 45 mg at Baseline.
- Ustekinumab 90 mg: Weeks 16-60: Adverse events which occurred during Weeks 16-60 in participants who were randomly assigned to ustekinumab 90 mg at Baseline.
Arm/Group | Placebo: Controlled Period | Ustekinumab 45 mg: Controlled Period | Ustekinumab 90 mg: Controlled Period | Placebo: Weeks 16-24 | Placebo -> Ustekinumab 45 mg: Weeks 16-60 | Ustekinumab 45 mg: Weeks 16-60 | Ustekinumab 90 mg: Weeks 16-60
Serious Adverse Events (participants affected / at risk) | 5/104 | 0/103 | 1/104 | 0/60 | 2/80 | 6/100 | 6/99
Other Adverse Events (participants affected / at risk) | 19/104 | 16/103 | 19/104 | 5/60 | 10/80 | 16/100 | 24/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Controlled Period (N=104) | Ustekinumab 45 mg: Controlled Period (N=103) | Ustekinumab 90 mg: Controlled Period (N=104) | Placebo: Weeks 16-24 (N=60) | Placebo -> Ustekinumab 45 mg: Weeks 16-60 (N=80) | Ustekinumab 45 mg: Weeks 16-60 (N=100) | Ustekinumab 90 mg: Weeks 16-60 (N=99)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular Insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Controlled Period (N=104) | Ustekinumab 45 mg: Controlled Period (N=103) | Ustekinumab 90 mg: Controlled Period (N=104) | Placebo: Weeks 16-24 (N=60) | Placebo -> Ustekinumab 45 mg: Weeks 16-60 (N=80) | Ustekinumab 45 mg: Weeks 16-60 (N=100) | Ustekinumab 90 mg: Weeks 16-60 (N=99)
Bronchitis (Infections and infestations) | 3 | 1 | 0 | 0 | 2 | 2 | 8
Nasopharyngitis (Infections and infestations) | 5 | 8 | 10 | 3 | 3 | 6 | 8
Sinusitis (Infections and infestations) | 3 | 1 | 3 | 0 | 1 | 0 | 5
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 1 | 1 | 6 | 2
Headache (Nervous system disorders) | 4 | 5 | 5 | 1 | 4 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.